CLINICAL TRIAL: NCT02805556
Title: Study of the Absolute Bioavailability of BMS-626529 in Healthy Subjects Following Oral Dosing of BMS-663068 and Intravenous Dosing of BMS-626529
Brief Title: Absolute Bioavailability of BMS-626529 After Oral and Intravenous Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206218; AI438-075 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2016-05-31; First posted 2016-06-20 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; BMS-626529

ARMS (1):
- Oral dose of BMS-663068 + intravenous dose of [13C]BMS 626529 (Experimental): Single oral dose of BMS-663068 followed by Single intravenous dose of [13C]BMS 626529
  Interventions: Drug: BMS-663068; Drug: BMS-626529

INTERVENTIONS:
Drug: BMS-663068 — Single oral dose of BMS-663068
Drug: BMS-626529 — Single intravenous dose of [13C]BMS 626529

SUMMARY:
A phase I absolute bioavailability study of BMS-626529 following oral and intravenous dosing

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* BMI 18.0-32.0 kg/m2
* Men sexually active with women of childbearing potential must follow instructions for contraception for the duration of treatment plus 90 days
* Men must refrain from sperm donation for the length of the study and for 90 days
* Sign informed consent

Exclusion Criteria:

* Significant medical illness
* Tobacco use in the last 12 months
* Major surgery within 4 weeks of study administration
* Donation of blood within 4 weeks of study administration
* Current or recent (within 3 months of study administration) of gastrointestinal disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
The absolute bioavailability of BMS-626529 after single oral (BMS-663068) and single intravenous dosing ([13C]-BMS-626529) by assessing the primary endpoints AUC(inf) | up to 11 days

SECONDARY OUTCOMES:
Safety and tolerability of single oral dose of BMS-663068 as determined by medical review of adverse event reports, vital sign measurements, electrocardiograms (ECGs), and results of physical examination and laboratory tests | up to 31 days
Safety and tolerability of single intravenous dose of [13C]-BMS-626529 as determined by medical review of adverse event reports, vital sign measurements, electrocardiograms (ECGs), and results of physical examination and laboratory tests | up to 31 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Lisburn, United Kingdom